CLINICAL TRIAL: NCT04551300
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Escalated and Fixed Doses of VS-505(AP301) in Comparison With Sevelamer Carbonate to Treat Hyperphosphatemia in Chronic Kidney Disease Patients Receiving Hemodialysis
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of VS-505(AP301) to Treat Hyperphosphatemia in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Alebund Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APCKD001
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Intervention Model Description: 4 different dosages of VS-505 in Comparison with Sevelamer Carbonate
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- VS-505 500mg (Experimental): VS-505 500mg (two 250 mg capsules) oral administration three times a day with meal, daily total dosage 1500mg.
  Interventions: Drug: VS-505
- VS-505 750mg (Experimental): VS-505 750mg (one 750 mg capsule) oral administration three times a day with meal, daily total dosage 2250mg.
  Interventions: Drug: VS-505
- VS-505 1500mg (Experimental): VS-505 1500mg (two 750 mg capsules) oral administration three times a day with meal, daily total dosage 4500mg.
  Interventions: Drug: VS-505
- VS-505 2250mg (Experimental): VS-505 2250mg (three 750 mg capsules) oral administration three times a day with meal, daily total dosage 6750mg.
  Interventions: Drug: VS-505
- Sevelamer Carbonate 1600mg (Active Comparator): Sevelamer Carbonate 1600mg (two 800mg pills) oral administration three times a day with meal, daily total dosage 4800mg.
  Interventions: Drug: Sevelamer Carbonate

INTERVENTIONS:
Drug: VS-505 — 4 dosages of experimental drug
  Arms: VS-505 1500mg; VS-505 2250mg; VS-505 500mg; VS-505 750mg
Drug: Sevelamer Carbonate — Active Comparator
  Other Names: Renvela
  Arms: Sevelamer Carbonate 1600mg

SUMMARY:
A multi-center, open-label, parallel-design, active-controlled phase 2 study to evaluate the tolerability, safety and efficacy of various dosages of VS-505 compared with Sevelamer Carbonate when given orally with meal for 6 weeks to treat hyperphosphatemia in chronic kidney disease subjects receiving maintenance hemodialysis.

DETAILED DESCRIPTION:
The main body of this study has 5 intervention arms, 4 VS-505 treatment arms of various dosage plus 1 active control arm of Sevelamer Carbonate, each consists 25 subjects. Prior to this main part, a dose escalating cohort of 25 subjects is added to evaluate the tolerability of VS-505 in Chinese patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults with end stage renal disease who are receiving a stable hemodialysis regimen (3 times per week) with sufficient dialysis adequacy;
* Serum phosphorus level range from >1.94 mmol/L (6.0 mg/dL) to ≤3.23 mmol/L (10.0 mg/dL) at the end of washout phase.

Exclusion Criteria:

* Kidney transplant patient or scheduled kidney transplant, or change to peritoneal dialysis, home hemodialysis or plan to relocate to another dialysis center during the study period；
* Serum phosphorus level is <1.29 mmol/L（4.0 mg/dL) or >2.42 mmol/L（7.5 mg/dL) at screening, or documented to be >3.23 mmol/L（10 mg/dL) within the latest three month prior to screening (screening included);
* Serum calcium level is <8 mg/dL or >11 mg/dL at the screening;
* Serum immunoreactive parathyroid hormone (iPTH)>1000 pg/mL at the screening;
* History of hemochromatosis or serum ferritin value ≥1000 μg/L at screening；
* Current clinically significant gastrointestinal (GI) disorder, or history of intestine obstruction, gastrectomy or duodenectomy, or GI tract surgery within 12 weeks prior to screening;
* Poorly controlled hypertension, cardiovascular disorders, and history of cerebrovascular disease or cardiovascular disease event within 24 weeks (6 months) prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus change from baseline to end of treatment | 6 weeks

SECONDARY OUTCOMES:
Time to serum phosphorus response，defined as serum phosphorus level decrease by 0.32 mmol/L（1 mg/dL）and serum phosphorus level below 1.78 mmol/L（5.5 mg/dL） | 6 weeks
The achievement rate of subjects with serum phosphorus in the target range 1.13-1.78 mmol/L（3.5-5.5 mg/dL）by the end of treatment | 6 weeks
Serum calcium change from baseline to end of treatment | 6 weeks
Serum Ca×P change from baseline to end of treatment | 6 weeks
Serum iPTH change from baseline to end of treatment | 6 weeks

OTHER OUTCOMES:
Serum ferritin change from baseline to end of treatment | 6 weeks
Number of serious adverse events (SAEs) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jilin Province People's Hospital, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Dalina Municipal Central Hospital, Dalian, Liaoning
  - The First Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong Universiity School of Medcine, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Zhuang B, Gan L, Liu B, Yuan W, Shi M, Peng A, Wang L, Chen X, Liu T, Zhang S, Wang S, Gao Q, Wang B, Zheng H, Liu C, Luo Y, Ye H, Lin H, Li Y, He Q, Zheng F, Luo P, Long G, Lu W, Li K, Yang J, Liu YC, Zhang Z, Li X, Zhang W, Zuo L. Tolerability, safety and efficacy of a novel phosphate binder VS-505 (AP301): a Phase 2 dose-escalation and dose-ranging study in patients undergoing maintenance hemodialysis. Nephrol Dial Transplant. 2024 Sep 27;39(10):1649-1661. doi: 10.1093/ndt/gfae053. PMID 38453435